CLINICAL TRIAL: NCT06067620
Title: Robotic Right Hemicolectomy With Intracorporeal Anastomosis Versus Laparoscopic Right Hemicolectomy With Extracorporeal Anastomosis (PRORHEM): a Randomized Controlled Trial
Brief Title: Robotic Right Hemicolectomy Versus Laparoscopic Right Hemicolectomy
Acronym: PRORHEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeremy Meyer (Other)
Collaborators: University Hospital, Geneva (Other); Spital Biel, Switzerland (Unknown); Hôpital Fribourgeois (Other)
Responsible Party: Sponsor-Investigator, Jeremy Meyer, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRORHEM
Record Dates: First submitted 2023-09-11; First posted 2023-10-05 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Neoplasms; Colorectal Neoplasms Malignant; Colorectal Neoplasms, Benign; Colorectal Cancer; Colorectal Polyp; Colorectal Adenoma; Colorectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic right hemicolectomy (Experimental): Robotic right hemicolectomy with intracorporeal anastomosis and extraction through a C-section (fully minimally invasive right hemicolectomy)
  Interventions: Procedure: Robotic right hemicolectomy
- Laparoscopic right hemicolectomy (Active Comparator): Laparoscopic right hemicolectomy with extracorporeal anastomosis and extraction through midline (standard of care)
  Interventions: Procedure: Laparoscopic right hemicolectomy

INTERVENTIONS:
Procedure: Robotic right hemicolectomy — Robotic right hemicolectomy with intracorporeal anastomosis and extraction through a C-section, using the Da Vinci Xi.
  Arms: Robotic right hemicolectomy
Procedure: Laparoscopic right hemicolectomy — Laparoscopic right hemicolectomy with extracorporeal anastomosis and extraction through midline.
  Arms: Laparoscopic right hemicolectomy

SUMMARY:
Robotic right hemicolectomy with intra-corporeal anastomosis may have better short-term recovery outcomes and decreased incidence of incisional hernia when compared to the laparoscopic actual standard of care, for similar safety outcomes.

DETAILED DESCRIPTION:
During laparoscopic right hemicolectomy (lapRHC) for cancer or polyp, intra-corporeal anastomosis (ICA) offers better short-term recovery and decreased incidence of incisional hernia (IH) when compared to extra-corporeal anastomosis (ECA). However, because of the technical limitations of laparoscopy, ICA has not gained in wide acceptance and ECA has remained the standard of care. On the contrary, robotics offers improved suturing capacities and facilitates the realization of ICA. Therefore, robotic right hemicolectomy (robRHC) with ICA may have better short-term recovery outcomes and decreased incidence of IH when compared to the laparoscopic actual standard of care. In a randomized controlled trial, we will compare robRHC with ICA with lapRHC with ECA, in terms of recovery of bowel function (time to first passage of faeces). Secondary outcomes will notably include length of stay, incidence of IH, patient-reported esthetical outcomes and safety outcomes (morbidity, mortality, proximal and distal margins, harvested lymph nodes).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring elective minimally invasive RHC for cT1-T3 Nx M0 cancer of the right colon (including cancer of the appendix, caecum, ascending colon and hepatic flexure).

Exclusion Criteria:

* Not scheduled for minimally invasive RHC (refuses surgery and/or planned open approach)
* Emergency surgery
* Hereditary colorectal cancer
* Inflammatory bowel disease
* Synchronous resection of (an)other organ(s)
* Synchronous surgical procedure (including more extended resection of the lower gastrointestinal tract)
* cT4
* cM+
* History of laparotomy
* Pregnancy
* No anastomosis planned
* Unable to provide informed consent
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first passage of faeces | From index surgical procedure (skin closure) until time of first passage of faeces, during hospitalisation, on average during the first 7 post-operative days
  Measured in hours, starting at the skin closure of the index surgery

SECONDARY OUTCOMES:
Duration of surgery | From skin incision to skin closure, during index surgical procedure
  Measured in minutes
Blood loss | From skin incision to skin closure, during index surgical procedure
  Measured in ml
Intra-operative transfusion | From skin incision to skin closure, during index surgical procedure
  Number of patients who received blood and/or blood products transfusion
Intra-operative complication | From skin incision to skin closure, during index surgical procedure
  Number of patients who experienced a complication during the index surgery
Conversion to open surgery | From skin incision to skin closure, during index surgical procedure
  Number of patients who had conversion to open surgery; defined as an extraction site longer than 10cm
Length of the extraction site | At post-operative day 30
  Measured in centimeters
Creation of a stoma | From skin incision to skin closure, during index surgical procedure
  Number of patients who received a stoma during the index surgery
Hb, WBC and CRP | At post-operative day 1, post-operative day 2, post-operative day 3, post-operative day 4 and post-operative day 5
  Blood tests
Time to first passage of flatus | From index surgical procedure (skin closure) until time of first passage of flatus, during hospitalisation, on average during the first 7 post-operative days
  Measured in hours, starting at the skin closure of the index surgery
In-hospital postoperative ileus | During hospitalisation, on average during the first 5 post-operative days
  Number of patients who experienced a post-operative ileus which required the insertion of a nasogastric tube
Length of stay | From the first day of hospitalisation to the day of discharge, on average during the first 10 post-operative days
  Measured in days
Post-operative morbidity | From index surgical procedure (skin closure) to post-operative day 30
  Number of patients who experienced post-operative morbidity, as measured by the Clavien-Dindo scale
Surgical site infection | From index surgical procedure (skin closure) to post-operative day 7 and post-operative day 30
  Number of patients who experienced surgical site infection
Anastomotic leak | From index surgical procedure (skin closure) to post-operative day 30
  Number of patients who experienced anastomotic leak, with radiological and/or surgical confirmation
Re-intervention | From index surgical procedure (skin closure) to post-operative day 30
  Number of patients who required a surgical re-intervention associated with the index surgery
Mortality | From index surgical procedure (skin closure) to post-operative day 30
  Number of patients who experienced mortality
Proximal margin | Within 10 days from the index surgical procedure
  Measured in centimeters, on the operative specimen of the index surgery
Distal margin | Within 10 days from the index surgical procedure
  Measured in centimeters, on the operative specimen of the index surgery
Harvested lymph nodes | Within 10 days from the index surgical procedure
  Number of harvested lymph nodes, on the operative specimen of the index surgery
Histology of the tumor/polyp | Within 10 days from the index surgical procedure
  Type of cancer and/or polyp, based on the operative specimen of the index surgery
TNM stage | Within 10 days from the index surgical procedure
  8th edition of the UICC TNM classification, based on the operative specimen of the index
Bowel function | At post-operative day 30 and post-operative year 1
  Gastrointestinal Quality of Life Index (GQLI)
Quality of recovery | At post-operative hour 12, post-operative day 1, post-operative day 2, post-operative day 3, post-operative day 4, post-operative day 5 and post-operative day 7
  Quality of Recovery-15 (QoR-15) score
Aesthetic numeric analogue scale (ANA-scale) | At post-operative day 30 and post-operative year 1
  Measuring the patient-reported esthetical aspect of the surgical wounds
Incidence of incisional hernia | At post-operative year 1
  Overall, and at extraction site; measured clinically and by CT

CONTACTS AND LOCATIONS:
Overall Officials: Christian Toso, MD, PhD, Study Chair — University Hospitals of Geneva

IPD SHARING:
Plan to Share IPD: No